CLINICAL TRIAL: NCT02175589
Title: Controlled Ceasing of Colchicine Therapy in Familial Mediterranean Fever (FMF) Patients With Single MEFV (Mediterranean Fever) Gene Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Schneider Children's Hospital (Other)
Responsible Party: Principal Investigator, yonatan butbul MD, Senior pediatrician & pediatric rheumatologist, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0080-14-RMB
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Familial Mediterranean Fever
Keywords: Familial Mediterranean Fever; Monozygous; MEFV; Colchicine; Serum Amyloid A
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Other): Colchicine Cessation in FMF patients with one MEFV mutation
  Interventions: Other: Colchicine Cessation
- Control group (No Intervention): The control group includes FMF patients that will be kept on a daily colchicine treatment

INTERVENTIONS:
Other: Colchicine Cessation — Colchicine Cessation
  Arms: Study group

SUMMARY:
The purpose of this study is to evaluate the effect of discontinuation of colchicine treatment in a specific group of asymptomatic FMF patients with a single mutation in MEFV gene, both from a clinical and laboratory aspects.

DETAILED DESCRIPTION:
The diagnosis of FMF is mainly clinical and genetic tests are only used to confirm the diagnosis . Even though the disease is autosomal recessive, not all FMF patients have two recognizable MEFV mutations. The phenotype of FMF patients varies according to the genotype, as shown by a number of studies showing that patients with one MEFV mutation have milder disease or even no symptoms. Some of the previously mentioned studies have shown that ceasing colchicine prophylaxis in these patients caused no recurrence. So far, no prospective controlled study has tested the effect of colchicine cessation in this group of FMF patients. The investigators presume that asymptomatic FMF patients with a single mutation can stop regular colchicine treatment while remaining under close follow-up.

The purpose of the work:

To examine the effect of colchicine cessation in a defined group of asymptomatic FMF patients with a single mutation in MEFV gene.

Methods and study population:

The work will be a controlled prospective comparative study including FMF patients aged 2-18 years. Patients included will be those who were asymptomatic for six months prior to entering the study and were regularly treated with colchicine, and with a normal serum level of Serum Amyloid A (SAA). The study group will include patients with a single MEFV mutation that will stop colchicine therapy, and the control group will include FMF who will continue regular colchicine treatment. Follow-up in both groups will include clinical and laboratory (serum SAA levels) evaluation.

The study end points and renewal of the colchicine:

Any patient that develops acute symptoms of FMF will be immediately invited to the rheumatology clinic for medical examination. In addition, patients will be invited to the clinic after 3 and 6 months from the beginning of the study. At any clinic visit (scheduled or not) the patients will be assessed clinically and laboratory (serum SAA levels). The study will be stopped and colchicine will be renewed if at any of the above mentioned clinic visit the patient will be diagnosed as having a classic FMF attack or the SAA level will be above 10 mg / l.

The importance of the study:

If the investigators conclude that colchicine prophylaxis can be safely discontinued in this group of FMF patients this will save them a treatment currently defined as a treatment for life.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with FMF based on clinical criteria
* FMF patients diagnosed of having at least one common MEFV mutation will be assigned to the study group. FMF patients who staid on colchicine treatment will be assigned to the control group, regardless of their genotype.
* Patients who were on a continuous colchicine prophylactic treatment for six months prior to entering the study.
* FMF patients who were free of acute FMF symptoms for six months prior to entering th study
* Patients were included in the study only if they had normal serum level of SAA (up to 10 mg / l).

Exclusion Criteria:

* Patients that in the six months prior to entering the study continued to have classic FMF episodes despite being on a continuous prophylactic colchicine
* Patients that had high level of SAA (above 10 mg/l) despite being on prophylactic colchicine treatment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Acute clinical episode of FMF | 6 months
  Acute clinical episode of FMF diagnosed by one of the investigators at any clinic visit assigned at 3 or 6 months after the cessation of colchicine treatment or at an unassigned visit if the patient attained the clinic due to an acute symptoms of FMF

SECONDARY OUTCOMES:
High level of Serum Amyloid A (SAA) in serum | 6 months
  High level of SAA (above 10 mg/l) at any clinic visit assigned at 3 or 6 months after the cessation of colchicine treatment or at an unassigned visit if the patient attained the clinic due to an acute symptoms of FMF

CONTACTS AND LOCATIONS:
Overall Officials: Yonatan Butbul, MD, Study Chair — Rambam Health Care Campus; Riva Brik, MD, Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Pediatric rheumatology clinic, Rambam Medical Center, Haifa
  - Schneider children's hospital, Petah Tikva